CLINICAL TRIAL: NCT00260676
Title: a Randomised Control Trial on Protective Ventilatory Strategy in Potential Organ Donors
Brief Title: Protective Ventilatory Strategy in Potential Organ Donors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Luciana Mascia, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 396
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Mechanical Ventilation
Keywords: brain death; lung transplantation; organ donors; potential organ donors
MeSH Terms: conditions — Brain Death

ARMS (1):
- conventional ventilation, protective ventilation (Other)
  Interventions: Procedure: change ventilation

INTERVENTIONS:
Procedure: change ventilation — reduction of tidal volume, increase of PEEP, recruiting maneuver, apnea test during CPAP

SUMMARY:
The aim of the study is to verify if a "PROTECTIVE" ventilatory strategy (low tidal volume and high PEEP, application of CPAP during the apnea test and recruitment maneuvers), improves lung function and increases the number of lungs eligible for transplantation.

DETAILED DESCRIPTION:
Lung transplantation reduces mortality in patients with severe pulmonary diseases. While 50-70% of kidney, liver and heart are eligible for transplantation, only 20% of the lungs fit the criteria for transplant. More than 30% of the lungs theoretically suitable for donation are not actually collected because following brain death they develop severe hypoxemia and abnormal chest X-ray. Guidelines for critical care management of potential organ donors suggest that after the diagnosis of brain death, treatment priority can be shifted from cerebral protection to a strategy aimed at preserving solid organ perfusion and function. However the ventilatory strategy recommended for potential lung donors is similar to the one proposed for brain injured patients. This ventilatory strategy based on high Vt and low PEEP may induce a further exacerbation of the pulmonary and systemic inflammatory response in patients with acute lung injury/acute respiratory distress syndrome. Moreover, recent data suggest that this strategy may be harmful in "normal lungs" of mechanical ventilated patients. Aim of the study is to verify if a "PROTECTIVE" ventilatory strategy (low tidal volume and high PEEP, application of CPAP during the apnea test and recruitment maneuvers) improves lung function. Primary end point of the study is to increase the number of lungs that meet the eligibility criteria for transplantation. Secondary end point is to increase the number of lungs really transplanted.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Chest X-ray: no infiltrates
* Duration of mechanical ventilation from the admission to ICU to the clinical diagnosis of brain death < 5 days
* No history of Smoking (1 pack/day for 20 years; 1/2 pack/day for 40 years; 2 packs/day for 10 years)
* No history of Asthma
* No history of COPD
* No history of Trauma
* No history of Thoracic surgery

Exclusion Criteria:

* Evidence of aspiration (chest X-ray or bronchoscopy) or sepsis
* Purulent secretions (tracheal suction or bronchoscopy)
* Sputum Gram stain with bacteria, fungus, significant number of WBC

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-09; Primary Completion 2009-09 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
To increase the number of lungs that meet the eligibility criteria for transplantation | end of brain death diagnosis observation period

SECONDARY OUTCOMES:
To increase the number of lungs really transplanted | end of brain death diagnosis observation period
Interim analysis at 100 subjects enrolled will be considered | six months after transplant

CONTACTS AND LOCATIONS:
Overall Officials: luciana mascia, MD PhD, Principal Investigator — University of Turin, Italy; marco ranieri, MD, Study Director — University of Turin, Italy
Locations (1):
- University of Turin, Department of Anesthesia and Intensive Care Medicine, Turin, Italy

REFERENCES:
- [Derived] Mascia L, Pasero D, Slutsky AS, Arguis MJ, Berardino M, Grasso S, Munari M, Boifava S, Cornara G, Della Corte F, Vivaldi N, Malacarne P, Del Gaudio P, Livigni S, Zavala E, Filippini C, Martin EL, Donadio PP, Mastromauro I, Ranieri VM. Effect of a lung protective strategy for organ donors on eligibility and availability of lungs for transplantation: a randomized controlled trial. JAMA. 2010 Dec 15;304(23):2620-7. doi: 10.1001/jama.2010.1796. PMID 21156950